CLINICAL TRIAL: NCT01325012
Title: Ultrasound-Guided Continuous Sciatic Nerve Blocks: Popliteal Versus Subgluteal Catheters
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Surgeon doing procedures amenable to this study left institution.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Subgluteal vs Popliteal
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Foot Surgery
Keywords: Pain; Surgery; Catheter; Nerve Block; Popliteal; Subgluteal; Sciatic; UCSD; Moderate-to-severe pain; Perineural Catheter; Orthopedic Surgery; foot surgery surgery; sciatic perineural catheter; age =>18
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subgluteal Sciatic Nerve Block (Active Comparator): Patients randomized to this group will receive a sciatic nerve block with the catheter tip insertion at the subgluteal location 1-3 cm caudad to the inferior border of the gluteus maximus muscle.
  Interventions: Procedure: Subgluteal Sciatic Nerve Block
- Popliteal Sciatic Nerve Block (Active Comparator): Patients randomized to this group will receive a sciatic nerve block with the catheter tip insertion at the popliteal location 1-3 cm cephalad to the sciatic bifurcation.
  Interventions: Procedure: Popliteal Sciatic Nerve Block

INTERVENTIONS:
Procedure: Subgluteal Sciatic Nerve Block — Patients randomized to this group will receive a sciatic nerve block with the catheter tip insertion at the subgluteal location 1-3 cm caudad to the inferior border of the gluteus maximus muscle. After catheter placement, outcome measures will be assessed.
  Arms: Subgluteal Sciatic Nerve Block
Procedure: Popliteal Sciatic Nerve Block — Patients randomized to this group will receive a sciatic nerve block with the catheter tip insertion at the popliteal location 1-3 cm cephalad to the sciatic bifurcation. After Catheter placement outcome measures will be assessed.
  Arms: Popliteal Sciatic Nerve Block

SUMMARY:
To determine the relationship between perineural catheter location along the sciatic nerve (popliteal versus subgluteal placement) and infusion effects for ultrasound-guided continuous sciatic nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* undergoing foot surgery with a sciatic perineural catheter for postoperative analgesia
* spending the first postoperative night hospitalized
* age 18 years or older

Exclusion Criteria:

* pregnancy
* inability to communicate with the investigators and hospital staff
* incarceration
* clinical neuropathy in the surgical extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Muscle Strength (MVIC) of the hamstring muscles | 08:00-09:00 morning after surgery as a percentage of baseline
  We will evaluate hamstring strength which is innervated by the sciatic nerve with an isometric force electromechanical dynamometer to measure the force produced during a maximum voluntary isometric contraction (MVIC) in a seated position with the knees flexed at 90º

SECONDARY OUTCOMES:
Sensory Effect | 08:00-09:00 morning after surgery
  We will evaluate tolerance of transcutaneous electrical stimulation. Electrocardiogram pads will be placed on the plantar and dorsal aspects of the foot, and attached to a nerve stimulator. The current will be increased from 0 mA until subjects described a "buzzing" sensation (not painful), at which time the current will be recorded as the tolerated level and the nerve stimulator turned off.
Pain Scores | from leaving the PACU until 08:00 the morning after surgery
  Surgical pain scores both average and worse as collected by nursing staff; and also the average and worse pain during the primary endpoint measurement
Sleep Disturbances | recorded at 08:00-09:00 the morning after surgery for the previous night
  Total number of times patient woke in the night due to surgical pain.
Total Infusion | recorded at 08:00-09:00 the morning following Surgery
  Total infusiond duration in time and volume and total number of boluses delivered via catheter.
Anesthetic Leakage | recorded at 08:00-09:00 the morning following Surgery
  Leakage from the catheter site noted by patient.
analgesic consumption | end of PACU stay until 08:00-09:00 the morning following surgery
  Hourly analgesic consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, Department of Anesthesiology
Locations (2):
- United States (2):
  - UCSD Medical Center, Thornton, La Jolla, California
  - UCSD Medical Center Hillcrest, San Diego, California